CLINICAL TRIAL: NCT05440825
Title: Self-management of Stress and Sleep Disturbances with Virtual Reality Relaxation for People with Burn-out, Mood, Anxiety or Psychotic Disorders: a Single-blind Randomized Controlled Trial
Brief Title: Self-management of Stress and Sleep Disturbances with Virtual Reality Relaxation
Acronym: Relax XL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Twente (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202100662
Record Dates: First submitted 2022-06-17; First posted 2022-07-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality
Keywords: virtual reality; relaxation; stress; sleep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VRelax (Experimental): Participants will be using Virtual Reality relaxation (VRelax) in addition to treatment as usual
  Interventions: Device: VRelax
- Relaxation exercises (Active Comparator): Participants will be using relaxation exercises in addition to treatment as usual
  Interventions: Other: Relaxation exercises

INTERVENTIONS:
Device: VRelax — Virtual Relaxation relaxation, VRelax, includes a collection of high quality 360° degrees videos of nature environments with 3D audio and interactive elements, created for relaxation, stress-reduction and improving sleep. When activated, the participant can choose specific 360° videos from a menu. The 360° videos include among other things a coral reef with an interactive game element of popping air bubbles, a scuba diving experience with dolphins, a mountain meadow with cows, and a session of Tibetan sound bowls.
  Arms: VRelax
Other: Relaxation exercises — Relaxation exercises consisting of audio-guided breathing exercises, muscle relaxation exercises, and body scan exercises
  Arms: Relaxation exercises

SUMMARY:
Stress is a well-established factor in the onset and continuation of burn-out anxiety, mood and psychotic disorders. Furthermore, sleep disturbances predispose and exacerbate mental health symptoms of the condition. In people with mental health problems, higher (social) stress-reactivity and impaired stress-recovery are present which is further aggravated by sleep disturbances and sleep deprivation. Relaxation reduces the stress, which in turn may reduce mental health symptoms, improve daily life functioning and quality of life. The burden of burn-out and psychiatric illness can be decreased by stress-reducing interventions which have been shown to improve quality of life and social and occupational functioning. Although current stress-reducing interventions appear to be efficacious, it must be taken into account that they require mental effort (i.e. attention and concentration of patients) which is often impaired in patients. To bridge this gap, a new e-Health application was developed called VRelax. VRelax is a virtual reality self-management stress-reduction tool (VRelax). This tool requires far less effort than traditional relaxation exercises due to its immersive properties, and has an immediate effect on perceived stress and emotional mental states. In this study, the short-, medium- and long term effect of VRelax + treatment as usual (TAU) compared to TAU and relaxation exercises on symptomatic recovery, level of social functioning, healthcare consumption and societal costs will be investigated.

DETAILED DESCRIPTION:
Once participants consent, they will complete the first assessment (T0). T0 starts with a physical assessment that consist of measuring weight, height, and waist circumference, a blood pressure test and a blood test. Furthermore, they will complete an assessment of physiological parameters during the use of VRelax. Then participants will complete a couple demographic questions, the Symptom Checklist-90-revised (SCL-90-R), the WHO Disability Assessment Schedule (WHO-DAS), the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST), the Hamilton Rating Scale for Depression (HRSD), and the Psychotic Symptom Rating Scales (Psyrats). Participants will then be informed to wear to different wearables for two weeks (Empatica E4 and MotionWatch 8). The instruction is to wear the Empatica E4 during the day to measure their Heart Rate (HR), Heart Rate Variability (HRV), and Skin Conductance (SC). The MotionWatch 8 will be worn during the night to measure their sleep. Participants also receive the instruction to complete the following online questionnaires at home: Burn-out Assessment Tool (BAT), Beck Anxiety Inventory (BAI), Inventory of Depressive Symptomatology Self Reported (IDS-SR), Mood Disorder Questionnaire (MDQ), Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI), Manchester Short Assessment of Quality of Life (MANSA), Recovery Assessment Scale - domains and stages (RAS-DS), Treatment Inventory of Costs in Patients (TiC-P), 36-item Short Form Survey (SF-36), and EQ-5D-5L.

Participants receive from their healthcare professional either VRelax or relaxation exercises with the instruction to use this for at least 20 minutes a day, at least five days a week, for six weeks. During those six weeks, participants will wear the wearables (Empatica E4 and MotionWatch 8) the first and the last week.

After six weeks after the first assessment, participants will complete the second assessment (T1). T1 is identical to T0 plus the System Usability Scale (SUS) for the participants who used VRelax. After 26 weeks after the first assessment, participants will complete the third assessment (T2). T2 consists of SCL-90-R, WHO-DAS, ASSIST, HRSD, Psyrats, BAT, BAI, IDS-SR, MDQ, PSS, PSQI, MANSA, TiC-P, SF-36, and EQ-5D-5L. The fourth and final assessment (T3) is 52 weeks after the first assessment. T3 is identical to T2.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment for burn-out, anxiety disorder, bipolar disorder, post-traumatic stress disorder, depressive disorder and/or psychotic disorder.
* Complaints of stress and/or sleep disturbances as reported by patient or therapist
* Age > 18

Exclusion Criteria:

* Individuals with a DSM-5 classification of substance use disorder
* Individuals with photosensitive epilepsy with seizure in the past year or organic brain damage
* Individuals with insufficient command of Dutch language
* Individuals with intellectual disability (estimated IQ < 70)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Checklist Scale - 90 - R | Between T0 and T1 (six weeks)
  The SCL-90-R is used to evaluate a broad range of psychological problems and symptoms of psychopathology during the last week.The SCL-90-R consists of 90 items scored on a five-point Likert scale.

SECONDARY OUTCOMES:
Changes in burn-out symptoms and stress | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The BAT is being used to evaluate the changes in burn-out symptoms and the PSS is being used to evaluate the changes in perceived stress. Both questionnaires have a five-point scale ranging from "never" to "always"
Changes in anxiety | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The BAI is is a self-report measure of anxiety. Each answer is being scored on a scale value of 0 (not at all) to 3 (severly). A higher total score indicate more severe anxiety
Changes in health and health-related quality of life | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The EQ-5D-5L is tool to measure health and health-related quality of life. The first 25 items of this questionnaires are based on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The patient is asked to indicate their health status by choosing the most appropriate level: no problems, slight problems, moderate problems, severe problems, and extreme problems. The last question is to indicate their current health status on a scale from 0 to 100.
Changes in depression | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The HRSD is a structured interview to assess the severity of depression. The HRSD contains 17 items pertaining to symptoms of depression experienced over the past week. The instruction for the researcher is to select the most appropriate answer which charaterizes the participant the best, ranging from "absent" to clearly present.
Changes in self-reported depressive symptoms | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The IDS-SR is a 3-item questionnaire measuring depressive symptoms. Each item has four statements that reflect various degrees of symptom severity, scored on a four-point scale from 0 to 3.
Changes in mood | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The MDQ is standard a 13-item self-report screening questionnaire with two optional questions that assesses symptoms of mania, hypomania, and depression. Participants check the "yes" or "no" boxes in response to answer. The second optional questions pertains to the level of functional impairment and has four answer options: no problem, minor problem, moderate problem, serious problem
Changes in psychotic symptoms | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The psyrats is a semi-structured interview to assess characteristics of hallucinations and delusions. The auditory hallucinations subscale (AHS) has 11 items. The delucions subscale (DS) has six items
Changes in psychosocial functioning | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The WHO-DAS II is an interview-administered 36-item questionnaire that covers six domains of functioning: cognition, mobility, self-care, getting along, life activities, participation. The participant is asked to indicate difficulties by selecting the most appropriate level: none, mild, moderate, severe, extreme or cannot do. In addition, the participant is asked on how many days these difficulties were present in the last 30 days: one day, less than a week, less than two weeks, more than two weeks, all days
Changes in quality of life | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The MANSA is a 16-item questionnaire to assess the quality of life. Satisfaction is rated on 7-point rating scale (1 = negative extreme, 7 = positive extreme)
Changes in recovery | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The Recovery Assessment Scale - Domains and Stages (RAS-DS) is a 38-item questionnaire to measure participants perceptions of individual recovery that they rate on a four-point scale: "untrue", "a bit untrue", "mostly true", "completely true"
Changes in substance use | Assessment at baseline, six weeks, 26 weeks, and 52 weeks
  The ASSIST is an 8-item interview that measures an participant's use of alcohol, tabacco products, and other drugss across his/her lifetime and in the past three months. The first item requires a "yes" or "no" answer while item 2 - 8 are scored on a five-point scale: never, once or twice, monthly, weekly, daily or almost daily
Change in sleep | Assessment at 26 weeks and 52 weeks
  The PSQI is a 19-item questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Each item is rated on a four-point scale: never, less than once a week, 1 - 2 times a week, 3 or more times a week
Change in medical use, medical cost and productivity losses | Assessment at 26 weeks and 52 weeks
  The TiC-P is a self-report questionnaire that consists of two parts. The first part includes 38 structured questions, starting with yes/no questions and followed by a question on the volume of medical consumption. The second part deals with questions about work.
Change in health-related quality of life | Assessment at 26 weeks and 52 weeks
  The SF-36 is a 36-item self-report questionnaire and measures eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Items are scored on different scales: yes/no scale, three-point scale, and five-point scale
Usability of VRelax | Assessment at 6 weeks
  The System Usability Scale (SUS) is being used to assess the usability of VRelax
24 h ambulatory measurement of electrodermal activity, cardiovascular activity, and sleep | The first and last week of using VRelax or relaxation exercises
  The MotionWatch 8 provides data on sleep (i.e. sleep latency, total sleep time, wake after sleep onset, sleep efficiency). The Empatica E4 provides data on electrodermal activity (Skin Conductance Level (SCL), number of Skin Conductance Responses (SCRs), Amplitude of the Skin conductance responses (S-AMPL)) and cardiovascular activity, time domain (mean RR interval, root mean square of successive differences between normal heartbeats (RMSSD), standard deviation of the normal sinus beats (SDNN))
Daily assessment of sleep | The first and last week of using VRelax or relaxation exercises
  A basic sleep diary that consist of questions about time of going to bed, time of falling asleep, time of waking up, and time of getting up
Daily pre- and post-session assessments of calness and relaxation | During the use of VRelax or relaxation exercises
  Within the VRelax environment, participants rate their level of calmness and relaxation with VAS items before and after each session. The group that is using the relaxation exercises, there is an online questionnaire to rate their pre- and post-session level of calmness and relaxation after using the relaxation exercises.
Changes in electodermal activity in laboratory setting | Assessment at baseline and six weeks
  The Shimmer 3 is being used to evaluate the electrodermal activity during the use of VRelax in laboratory setting
Changes in cardiovascular activity in laboratory setting | Assessment at baseline and six weeks
  The Shimmer 3 is being used to evaluate the cardiovascular activity during the use of VRelax in laboratory setting
Changes in physiological markers for comorbid somatic disease - weight | Assessment at baseline and six weeks
  A scale is being used to evaluate changes in weight
Changes in physiological markers for comorbid somatic disease - height | Assessment at baseline and six weeks
  A measurement tape is being used to evaluate changes in height
Changes in physiological markers for comorbid somatic disease - waist circumference | Assessment at baseline and six weeks
  A measurement tape is being used to evaluate changes in waist circumference
Changes in physiological markers for comorbid somatic disease - blood pressure | Assessment at baseline and six weeks
  A blood pressure monitor is being used to evaluate changes in blood pressure
Changes in physiological markers for comorbid somatic disease - blood | Assessment at baseline and six weeks
  Blood is being drawn to evaluate the changes in HBA1c, glucose, TC, HDL-C, TC-HDC-ratio, LDL-c, triglyceriden, creatinine (eGFR)

CONTACTS AND LOCATIONS:
Overall Officials: Catheleine van Driel, Principal Investigator — University Medical Center Groningen; Wim Veling, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Mediant, Enschede
  - Forte GGZ, Groningen
  - Lentis, Groningen
  - UMCG, Groningen
  - Argo GGZ, Lochem

IPD SHARING:
Plan to Share IPD: No